CLINICAL TRIAL: NCT07278271
Title: Toma de Decisiones en la Admisión Hospitalaria al Parto Con Ecografía Transperineal vs. Tacto Vaginal: Estudio Aleatorizado Controlado
Brief Title: Decision-Making in Labor Admission Using Transperineal Ultrasound vs. Vaginal Examination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Marcos Javier Cuerva González, Attending Obstetrician and Principal Investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI-4053
Record Dates: First submitted 2025-05-07; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Labor Active Dilated Cm
Keywords: Transperineal ultrasound; Intrapartum ultrasound; Vaginal examination; Hospital admission in labor; Term pregnancy; Angle of progression; Cervical dilatation; Ultrasound vs vaginal exam
MeSH Terms: interventions — Gynecological Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transperineal Ultrasound (Experimental): Participants in this arm will undergo transperineal ultrasound to assess cervical dilatation, angle of progression (AOP), fetal head position, and head-perineum distance (HPD). Hospital admission will be based on predefined sonographic criteria (e.g., dilation ≥3 cm or angle of progression >120° plus regular uterine contractions).
  Interventions: Diagnostic Test: Transperineal Ultrasound
- Vaginal Examination (Active Comparator): Participants in this arm will undergo standard digital vaginal examination. Hospital admission will be based on cervical dilation ≥4 cm and regular uterine contractions, following the routine clinical protocol.
  Interventions: Diagnostic Test: Vaginal Examination

INTERVENTIONS:
Diagnostic Test: Transperineal Ultrasound — Transperineal ultrasound will be performed to assess cervical dilatation, angle of progression, fetal head position, and head-perineum distance. Admission decisions will be made based on predefined sonographic thresholds.
  Arms: Transperineal Ultrasound
Diagnostic Test: Vaginal Examination — Standard digital vaginal examination will be conducted to assess cervical dilatation. Admission decisions will follow institutional protocol (≥4 cm dilation with regular contractions).
  Arms: Vaginal Examination

SUMMARY:
This clinical trial aims to determine whether transperineal ultrasound (a perineal external scan) can improve decision-making for hospital admission in term pregnant women in labor compared to traditional vaginal examination. Term pregnant women (>37 weeks) presenting with contractions at the emergency department will be randomly assigned to undergo either a transperineal ultrasound or a vaginal examination upon arrival. The study will evaluate whether ultrasound-based assessment reduces the rate of labor inductions and decreases patient discomfort during the admission evaluation. All participants will receive standard clinical evaluation and follow-up according to the assigned method, report discomfort levels using a standardized scale, and have labor outcomes recorded - including induction, oxytocin use, time to delivery, and mode of delivery -, to determine whether ultrasound improves clinical decision-making and maternal comfort.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled clinical trial is designed to evaluate whether transperineal ultrasound provides a more effective and less discomforting method than standard vaginal examination for decision-making regarding hospital admission in term pregnant women presenting with contractions. Vaginal examination remains the standard approach for assessing labor progression but is known to be subjective, poorly reproducible, and frequently uncomfortable for patients. In contrast, transperineal ultrasound offers objective and reproducible parameters such as cervical dilation, fetal head station, angle of progression, and head-perineum distance. Incorporating these measurements into the clinical evaluation may optimize admission criteria, reduce unnecessary hospitalizations, and lower the rate of labor inductions. After obtaining informed consent, eligible participants will be randomly assigned in a 1:1 ratio to either a transperineal ultrasound group or a standard vaginal examination group. In the ultrasound group, hospital admission will be recommended when cervical dilation is ≥3 cm or the angle of progression exceeds 120°, in the presence of regular uterine contractions. In the vaginal examination group, admission will be recommended when cervical dilation is ≥4 cm with regular contractions. Maternal discomfort during the evaluation will be assessed on a 0-10 numerical scale, and all labor outcomes and interventions will be recorded in standardized case report forms. A total of 170 participants (85 per group) will be enrolled to detect an 18% difference in labor induction rates with 80% power and a 95% confidence level. Statistical analyses will include descriptive and comparative methods (Chi-square, t-test, or non-parametric equivalents), with significance defined as p<0.05. The study will adhere to the principles of the Declaration of Helsinki and comply with applicable data protection regulations, including the Spanish Ley Orgánica de Protección de Datos (Organic Law on Data Protection, LOPD) and the European General Data Protection Regulation (GDPR).All participants will provide written informed consent prior to inclusion, and all data will be anonymized. The protocol has received approval from the institutional ethics committee. This trial builds upon prior observational findings demonstrating high agreement between ultrasound-based and traditional methods for assessing labor progression. By generating high-level evidence, it aims to support the implementation of transperineal ultrasound in labor triage protocols, improving the accuracy of clinical decision-making, enhancing maternal comfort, and contributing to better obstetric outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45 years
* Singleton pregnancy
* Gestational age ≥ 37 weeks (term pregnancy)
* Spontaneous uterine contractions at the time of presentation to the emergency department
* Cephalic presentation
* Willingness and ability to provide written informed consent

Exclusion Criteria:

* Premature rupture of membranes (PROM)
* Multiple gestation
* Known high-risk pregnancy (e.g., preeclampsia, intrauterine growth restriction, insulin-dependent diabetes)
* Previous cesarean delivery
* Breech or other non-cephalic presentation
* Elective cesarean section planned or requested
* Refusal to undergo vaginal delivery
* Inability or unwillingness to comply with the study protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility to participate in this study is based on biological sex, as only individuals who are biologically female can become pregnant and experience labor.
Enrollment: 170 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Labor Induction | From hospital admission decision to delivery
  Proportion of participants who undergo labor induction if admitted after evaluation by transperineal ultrasound or vaginal examination.

SECONDARY OUTCOMES:
Use of Oxytocin for Labor Augmentation | During labor (up to delivery)
  Proportion of participants who receive oxytocin for augmentation of labor following initial triage evaluation.
Time from Admission to Delivery | From hospital admission to time of delivery
Mode of Delivery (as recorded in the medical record) | At birth
  Mode of delivery will be recorded from the medical record and categorized as spontaneous vaginal delivery, assisted vaginal delivery (instrumental), or cesarean section.
Number of Vaginal Examinations Performed | From hospital admission for labor to delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study (after de-identification) will be made available to researchers upon reasonable request. This will include data on primary and secondary outcomes. Data will be shared after publication of the main results and with approval from the principal investigator and institutional ethics committee. Requests should be directed to Dr. Marcos J. Cuerva at marcosj.cuerva@salud.madrid.org

REFERENCES:
- [Background] Cuerva MJ, Garcia-Casarrubios P, Garcia-Calvo L, Gutierrez-Simon M, Ordas P, Magdaleno F, Bartha JL; ITU-R12 Group. Use of intrapartum ultrasound in term pregnant women with contractions before hospital admission. Acta Obstet Gynecol Scand. 2019 Feb;98(2):162-166. doi: 10.1111/aogs.13474. Epub 2018 Oct 30. PMID 30288731